CLINICAL TRIAL: NCT04935619
Title: Effects of Extended Cannabis Abstinence on Clinical and Cognitive Outcomes in Patients With Co-Morbid Major Depressive and Cannabis Use Disorders
Brief Title: Extended Effects of Cannabis Abstinence on Clinical Symptoms and Cognition in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 125-2020
Record Dates: First submitted 2021-06-01; First posted 2021-06-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cannabis Use; Major Depressive Disorder; Cognitive Impairment
Keywords: cannabis; substance abuse; depression; anxiety; contingency reinforcement
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction; Marijuana Abuse; Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Contingency Reinforcement Group (Other): Subjects assigned to the NCR group with self-reported abstinence verified by urinary THC-COOH level <20 ng/ml will not receive contingency monetary reinforcement at Day 28 of the study.
  Interventions: Behavioral: Non-Contingency Reinforcement
- Contingency Reinforcement Group (Experimental): Subjects assigned to the CR group with self-reported abstinence verified by urinary THC-COOH level <20 ng/ml will receive contingency monetary reinforcement at Day 28 of the study.
  Interventions: Behavioral: Contingency Reinforcement

INTERVENTIONS:
Behavioral: Contingency Reinforcement — Subjects will be randomly assigned on a 1:1 ratio to either the Contingency Reinforcement or Non-Contingency Reinforcement Intervention prior to their in-person screening visit.
  Arms: Contingency Reinforcement Group
Behavioral: Non-Contingency Reinforcement — Subjects will be randomly assigned on a 1:1 ratio to either the Contingency Reinforcement or Non-Contingency Reinforcement Intervention prior to their in-person screening visit.
  Arms: Non-Contingency Reinforcement Group

SUMMARY:
The prevalence of major depressive disorder (MDD) is ~5.0%, and rates of co-occurring SUDs in these patients approach 40-50%. Specifically, rates of co-morbid cannabis use disorder (CUD) in patients with MDD are elevated 2-3 fold compared to 2.9% in the general population, and is associated with poorer treatment outcomes and impaired cognitive and psychosocial functioning in comparison to MDD patients without CUD. Most studies of cannabis use in MDD are cross-sectional in design, and therefore causal relationships are unclear. This study investigates the effects of cannabis abstinence over a 28-day period in patients with MDD with co-occurring CUD using a randomized controlled design, namely contingent reinforcement.

DETAILED DESCRIPTION:
The prevalence of major depressive disorder (MDD) is ~5.0%, and rates of co-occurring SUDs in these patients approach 40-50%. Specifically, rates of co-morbid cannabis use disorder (CUD) in patients with MDD are elevated 2-3 fold compared to 2.9% in the general population, and is associated with poorer treatment outcomes and impaired cognitive and psychosocial functioning in comparison to MDD patients without CUD. To date, most studies of cannabis use in MDD were cross-sectional in design, and therefore causal relationships are unclear. The investigators previous studies in cannabis dependent patients with schizophrenia suggest that extended cannabis abstinence (up to 28 days) using contingent reinforcement is associated with improvements in specific areas of cognition (e.g. verbal learning and memory) and depressive symptoms. A more recent study using an open-label design demonstrated that 28 days of cannabis abstinence improves depressive symptoms and anhedonia in participants (N=11) with co-occurring MDD and CUD.

The investigators propose a controlled cannabis abstinence paradigm in patients with co-morbid MDD and CUD (N=52) to further investigate these findings. Stabilized MDD patients with moderate to severe CUD will be randomly assigned to one of two groups: 1) A contingent reinforcement (CR) intervention (n=26); 2) a non-contingent reinforcement (NCR) intervention (n=26), which will serve as a time and non-abstinence control. In the CR group, subjects achieving biochemically-verified cannabis abstinence at study endpoint (Day 28) will receive a $300 contingent payment; participants in the NCR group will not receive this contingent payment. The primary outcomes are: 1) cannabis abstinence rates at Day 28 in CR versus NCR groups; 2) changes in mood (depressive), anxiety and sleep symptoms over the 28-day assessment period. Secondary outcomes include cognition.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be between the ages 18-55
* Meet SCID for DSM-5 diagnostic criteria for cannabis use disorder, moderate to severe
* Meet SCID for DSM-5 diagnostic criteria for Major Depressive Disorder
* Be an outpatient receiving a stable dose of antidepressant medication for at least three months (to ensure stability of depressive symptoms
* Have a Hamilton Depression Rating Scale (HDRS-17) at baseline assessment in the range of 12-25..
* Have a Full-Scale IQ ≥ 80 as determined by the WTAR
* Be a non-treatment seeking cannabis user
* Evidence of sufficient motivation and effort as measured by a Test of Memory Malingering (TOMM) score ≥ 45.

Exclusion Criteria:

* Meets criteria for substance use disorder of alcohol or other illicit substances within the past 6 months (with the exception of cannabis, nicotine, or caffeine)
* Positive urine screen for illicit substances other than cannabis, nicotine, or caffeine
* Current suicidal or homicidal ideation
* Psychotic disorder diagnosis (e.g. schizoaffective disorder, major depression with psychotic features) as determined by the SCID
* Treatment seeking for cannabis use
* Meet SCID for DSM-5 diagnostic criteria for Bipolar Disorder
* Head Injury> 5 minutes LOC
* Exceed upper and lower cut-offs on HSRD-17 (See Inclusion Criteria)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Depressive Symptomology from Baseline to Week 4 | [Time Frame: Weekly (Day 0, Day 7, Day 14, Day 21, Day 28)]
  The Hamilton Depression Rating Scale will be administered to assess severity of depressive symptoms. [Min score = 0, Max score = 52; Higher scores evince more severe symptomology]
Changes in Anxious Symptomology from Baseline to Week 4 | [Time Frame: Weekly (Day 0, Day 7, Day 14, Day 21, Day 28)]
  The Beck Anxiety Inventory will be administered to assess severity of anxiety symptoms [Min score = 0, Max score = 63; Higher scores evince more severe symptomology].
Changes in Sleep Symptomology from Baseline to Week 4 | [Time Frame: Weekly (Day 0, Day 7, Day 14, Day 21, Day 28)]
  The Pittsburgh Sleep Quality Index will be administered weekly to examine quality of sleep and other sleep disturbances [Min score = 0, Max score = 21; Higher scores evince more severe symptomology].
Changes in Anhedonia from Baseline to Week 4 | [Time Frame: Weekly (Day 0, Day 7, Day 14, Day 21, Day 28)]
  The Snaith-Hamilton Pleasure Scale will be administered weekly to measure changes in anhedonia [Min score = 0, Max score = 14; Higher scores evince more severe symptomology].

SECONDARY OUTCOMES:
Changes in Verbal Learning and Memory | Day 0 and Day 28
  The Hopkins Verbal Learning Test will be administered to investigate this cognitive domain.
Changes in Attention and Visual Search | Day 0 and Day 28
  The Trail Making Test will be administered to investigate these cognitive domains
Changes in Working Memory | Day 0 and Day 28
  The Digit Span test will be administered to investigate this cognitive domain.
Changes in Sustained Attention | Day 0 and Day 28
  The Continuous Performance Test will be administered to investigate this cognitive domain

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, MD., FRCPC, Principal Investigator — CAMH
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No